CLINICAL TRIAL: NCT06687512
Title: An Exploratory, Proof-of-Concept, Double-Blind, Placebo-Controlled, Randomized, Comparative, Interventional, Prospective, Safety In-Use Tolerability and Efficacy Study of Test Products in Patients With Mild to Moderate Atopic Dermatitis (AD).
Brief Title: A Clinical Study to Assess the Safety and Effectiveness of Test Products in Mild to Moderate Atopic Dermatitis (AD) Patients.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Blossom Microbiotics LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NB240037-BM
Record Dates: First submitted 2024-10-19; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-Blind Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SaaTwae Bio-Natural Moisturizing Cream (Experimental): Mode of Usage: Apply a generous amount of the test product to the affected areas of atopic dermatitis. Gently massage the product into the skin until fully absorbed. Ensure that the application is consistent, especially after bathing or during flare-ups.
  Frequency: Twice a day (Once before going to the bed and once after bathing and drying off and during flare ups/itching) Route of Administration: Topical
  Interventions: Other: SaaTwae Bio-Natural Moisturizing Cream
- Placebo (Placebo Comparator): Mode of Usage: Apply a generous amount of the test product to the affected areas of atopic dermatitis. Gently massage the product into the skin until fully absorbed. Ensure that the application is consistent, especially after bathing or during flare-ups.
  Frequency: Twice a day (Once before going to the bed and once after bathing and drying off and during flare ups/itching) Route of Administration: Topical
  Interventions: Other: Placebo

INTERVENTIONS:
Other: SaaTwae Bio-Natural Moisturizing Cream — Mode of Usage: Apply a generous amount of the test product to the affected areas of atopic dermatitis. Gently massage the product into the skin until fully absorbed. Ensure that the application is consistent, especially after bathing or during flare-ups.
  Frequency: Twice a day (Once before going to the bed and once after bathing and drying off and during flare ups/itching) Route of Administration: Topical
  Arms: SaaTwae Bio-Natural Moisturizing Cream
Other: Placebo — Mode of Usage: Apply a generous amount of the test product to the affected areas of atopic dermatitis. Gently massage the product into the skin until fully absorbed. Ensure that the application is consistent, especially after bathing or during flare-ups.
  Frequency: Twice a day (Once before going to the bed and once after bathing and drying off and during flare ups/itching) Route of Administration: Topical
  Arms: Placebo

SUMMARY:
This is an exploratory, proof-of-concept, double-blind, placebo-controlled, randomized, comparative, interventional, prospective, safety in-use tolerability and efficacy study of test products in patients with mild to moderate Atopic Dermatitis.

DETAILED DESCRIPTION:
A total of 44 patients with mild to moderate Atopic Dermatitis for at least 6 months will be enrolled in the study to complete 40 patients having confirmed diagnosis of atopic dermatitis.

Subjects will be pre-screened by the screening department of NovoBliss Research. Subjects will be called on the telephone by the recruiting department.

A sufficient number of patients and children patients with legal parent or legal guardian will be pre-screened based on the moisture level by Corneometer® CM 825 and trans epidermal water loss by TEWAMeter® TM Hex followed by photographic collection of the active site for atopic dermatitis to ensure that enough subjects successfully qualify for screening before EC approval. The potential subjects will be screened as per the inclusion & exclusion criteria only after obtaining written informed consent from the subjects.

The subjects will be instructed to visit the facility as per the below visits. Visit 01 (Day 01): Screening, Randomization, Baseline Evaluation, Post application evaluation Visit 02 (Day 15 ±2 Days): Test products usage, Telephonic Follow-up Visit 03 (Day 30 ±2 Days): Test products usage, Evaluations. Visit 04 (Day 60 ±2 Days): Final Evaluation, End of Study.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age: For children: 6 years and above (both inclusive) at the time of parental consent/assent and For Adults: 18 to 65 years (both inclusive) at the time of consent.

  2) Sex: Healthy children (male or female) and adults (males and non-pregnant/non-lactating females) with mild to moderate atopic dermatitis.

  3) Subject's with TEWL >15% and Moisture level <20% at the time of screening. 4) Subject's with mild to moderate Atopic Dermatitis determined by Eczema Area and Severity Index (EASI) score with moderate erythema (redness: score 2) and mild scratch mark (scratching: score 1) will be enrolled into the study.

  5) Subject is diagnosed with mild to moderate atopic dermatitis with at least 1 active lesion that are accessible for instrumental measurements.

  6) Females of childbearing potential should have a negative urine pregnancy test at the time of screening visit.

  7) Subjects (adults and children) are generally in good general health as determined from a recent medical history, except for the atopic dermatitis.

  8) If subjects (adults and children) are using or taking any prescription or over the counter (OTC) medications prescribed by their physicians, they must be taking the medication for at least 4 weeks.

  9) Subject's and child's legal parent or guardian must agree to use the same brands and agree not to switch brands or variants of any skin care products during the study period.

  10) Subject's and child's legal parent or guardian must agree to limit the sun exposure to affected areas such as arms, legs covered during prolonged sun exposure.

  11) Subject's and child's legal parent or guardian must agree to dress the subjects in loose clothing to allow easy exposure to the entire body during study visits and throughout study duration of 60 days.

  12) Subjects and Legal parent or guardian must avoid allowing the subject a hot or cold beverage within one hour of their scheduled visits and for the duration of all clinic visits, warm beverages are allowed.

  13) Subjects and Legal parent or guardian must avoid allowing subject to swim or play in chlorinated water during study period.

  14) Subjects are not allowed to participate in any other study until this study is complete.

  15) Subjects and child's legal parent or guardian must be willing and able to follow the study directions and to return for all specified visits with the subject.

  16) Subjects and Child's legal parent or guardian must be willing to stop using all of the subject's normal body lotions for the duration of the study (8 weeks) and to use the provided test daily lotion as directed.

  17) Subjects and Child's legal parent or guardian must agree to record each use of the test products in the subject's diary card on daily basis.

  18) Subjects and Child's legal parent or guardian must agree to record medication use during the study.

  19) Subject's and child's legal parent or guardian must read, sign, and receive a copy of Informed Consent/Parental Informed Consent prior to initiate of study procedures.

  20) Having childbearing potential, is practicing and agrees to maintain an established method of birth control (IUD, hormonal implant device/injection, regular use of birth control pills or patch, diaphragm, condoms with spermicide or sponge with spermicidal jelly, cream or foam, partner vasectomy or abstinence). Females will be considered as non-childbearing potential if they are surgically sterile, have been post-menopausal for at least 1 year or have had a tubal ligation.

  21) Subjects willing to give written informed consent and are willing to come for regular follow up.

  22) Subjects have not participated in a similar investigation in the past three months.

  23) Subjects willing to use test product throughout the study period.

Exclusion Criteria:

* 1)Subjects with AD on the scalp (with hair), palms, and soles. 2) Subjects with active skin infections. 3) Subjects with other dermatologic diseases besides AD whose presence or treatments could interfere with the assessment of disease (eg, Psoriasis).

  4) Subjects who used systemic immunosuppressants within 4 weeks, topical steroids or immunomodulators within 1 week, moisturizers within 12 hours before evaluation.

  5) Subjects with milk allergies. 6) Change in current prescriptions (within 4 weeks of screening) or new and/or additional prescriptions for the skin condition (within 4 weeks of screening) or during the study.

  7) The subject has a known allergy or sensitivity to soaps, lotions, detergents, detanglers or fragrances.

  8) The subject has any other skin conditions i.e. cuts, scratches, ring worms, etc. which in the opinion of the Investigator, will interfere with the study results or will create undue risk for the subject.

  9) The subject has any of the conditions or factors that the Investigator believes may affect the response of the skin or the interpretation of the test results.

  10) Subjects having diabetes, hepatitis, epilepsy, thyroid or have or had any kind of cancer.

  11) The subject is currently taking or has taken any medication, which the Investigator believes may influence the interpretation of the data, such as 3 or more dosage or 3 or more days of anti-inflammatories (within 1 week of study enrolment) or anti-histamines and steroids.

  12) The subject must not have participated in a clinical study within 4 weeks prior to the screening visit of this study.

  13) Any other condition which could warrant exclusion from the study, as per the dermatologist's/investigator's discretion.

  14) Pregnant or breastfeeding or planning to become pregnant during the study period.

  15) History of chronic illness which may influence the cutaneous state.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2025-02-20 (Estimated); Study Completion 2025-02-20 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effectiveness of the test products in terms of change in Dry Skin/Ichthyosis Area and Severity Index (DASI) | baseline before usage on Day 01 and after usage of the test products at T30 minutes on Day 01, Day 30 (±2 Days) and Day 60 (±2 Days)
  Scale indicates 0-4 categorical scale (0: absent, 1: slight, 2: moderate, 3: severe, 4: extreme)
To evaluate the effectiveness of the test products in terms of changes in SCORAD severity scoring, | before usage of the test products on Day 01 and after usage of test products at T30 mins on Day 01, Day 30 (± 2 Days), Day 60 (± 2 Days).
  Scoring scale indicates 1 indicates mild intensity, 2 indicates moderate intensity, and 3 indicates severe intensity
To evaluate the effectiveness of the test products in terms of changes in Eczema Area and Severity Index | before usage of the test products on Day 01 and after usage of test products at T30 minutes on Day 01, Day 30 (± 2 Days), Day 60 (± 2 Days).
  Scoring Scale indicates none (0), mild (1), moderate (2) and severe (3).
To evaluate the effectiveness of the test products in terms of changes in visual assessment of post inflammatory hyperpigmentation | before usage of the test products on Day 01 and after usage of test products at T30 minutes on Day 01, Day 30 (± 2 Days), Day 60 (± 2 Days).
  Scoring scale indicates a 0-4 categorical scale (0: absent, 1: slight, 2: mild, 3: moderate, 4: maximum)

SECONDARY OUTCOMES:
To evaluate the effectiveness of the test products in terms of changes in visual and tactile assessment of skin scaliness | before usage of the test products on Day 01 and after usage of test products at T30 minutes on Day 01, Day 30 (± 2 Days), Day 60 (± 2 Days).
  Scoring scale indicates 0: absent and 4: extreme
To evaluate the effectiveness of the test products in terms of changes in visual and tactile | before usage of the test products on Day 01 and after usage of test products at T30 minutes on Day 01, Day 30 (± 2 Days), Day 60 (± 2 Days).
  Scoring scale indicates 0: absent and 4: extreme
To evaluate the effectiveness of the test products in terms of changes in visual and tactile assessment of skin redness | before usage of the test products on Day 01 and after usage of test products at T30 minutes on Day 01, Day 30 (± 2 Days), Day 60 (± 2 Days).
  Scoring scale indicates 0: absent and 4: extreme
To evaluate the effectiveness of the test products in terms of changes in visual and tactile assessment of skin itchiness | before usage of the test products on Day 01 and after usage of test products at T30 minutes on Day 01, Day 30 (± 2 Days), Day 60 (± 2 Days).
  Scoring scale indicates 0: absent and 4: Severe
To evaluate the effectiveness of the test products in terms of changes in visual and tactile assessment of skin dryness | before usage of the test products on Day 01 and after usage of test products at T30 minutes on Day 01, Day 30 (± 2 Days), Day 60 (± 2 Days).
  Scoring scale indicates 0: absent and 4: Severe
To evaluate the effectiveness of the test products in terms of changes in visual and tactile assessment of skin smoothness | before usage of the test products on Day 01 and after usage of test products at T30 minutes on Day 01, Day 30 (± 2 Days), Day 60 (± 2 Days).
  Scoring scale indicates 0: absent and 4: Severe
To evaluate the effectiveness of the test products in terms of changes in Visual Analogue Scale for Itching | before usage of the test products on Day 01 and after usage of test products at T30 minutes on Day 01, Day 30 (± 2 Days), Day 60 (± 2 Days).
  Scale where 0 indicates No itching and 100 indicates most severe itching imaginable
To evaluate the effectiveness of the test products in terms of changes in skin hydration | baseline before usage and after usage of the test products at T30 minutes on Day 01, Day 30 (±2 Days) and Day 60 (±2 Days)
  Change in skin hydration by Corneometer CM 825
To evaluate the effectiveness of the test products in terms of changes in skin barrier function | before usage and after usage of the test products at T30 minutes on Day 01, Day 30 (±2 Days) and Day 60 (±2 Days)
  Change in skin barrier function using TEWAMeter TM Hex
To evaluate the effectiveness of the test products in terms of changes in skin topography | before usage and after usage of the test products at T30 minutes on Day 01, Day 30 (±2 Days) and Day 60 (±2 Days)
  Change in skin topography by VISIOSCAN VC 20
To evaluate the effectiveness impact of the test products in the shift of skin microbiome by collecting skin swab | before usage and after usage of the test products at T30 minutes on Day 01, Day 30 (±2 Days) and Day 60 (±2 Days)
  Change in shift of skin microbiome by collection skin swab.
To evaluate the effectiveness of the test products in terms of changes in product perception questionnaire | before usage and after usage of the test products at T30 minutes on Day 01, Day 30 (±2 Days) and Day 60 (±2 Days)
  Questionnaire scale indicates 1: Not at all and 5: to large extent

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nayan K Patel, Principal Investigator — NovoBliss Research Pvt Ltd

IPD SHARING:
Plan to Share IPD: No